CLINICAL TRIAL: NCT07390201
Title: Effect of Sensory Integration Therapy on Gait Variability and Quality Of Life in Patients With Multiple Sclerosis: A Randomized Controlled Trial
Brief Title: Effect of Sensory Integration Therapy on Gait Variability and Quality Of Life in Patients With Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Mohamed Gamal Mahrous, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005138
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physical therapy program (Active Comparator): The Patients in this group will be treated by the conventional physical therapy program, two times a week for eight successive weeks (16 sessions in total for 70 min and enough rest in between).
  Interventions: Other: Conventional physical therapy program
- Conventional physical therapy program + Sensory integration therapy (Experimental): Patients in this group will be treated by the same conventional physical therapy program (30 min), in addition to sensory integration therapy program (SIT) (40 min). The most commonly duration and frequency of sessions will be 70 min and (16 treatment sessions for two times a week) for eight successive weeks.
  Interventions: Other: Conventional physical therapy program; Other: Sensory integration therapy

INTERVENTIONS:
Other: Conventional physical therapy program — This group will undergo a conventional physical therapy program twice weekly for eight weeks (16 sessions), with each 70-minute session including rest as needed. Sessions consist of a 5-minute warm-up, an active phase with individualized moderate-intensity aerobic exercises (64-76% of maximum heart rate) such as marching and over-ground walking with progressive difficulty, along with lower-limb stretching and strengthening exercises. Each session ends with a 5-minute cool-down using gentle stretching or gradual reduction of activity to minimize stiffness and muscle soreness.
Other: Sensory integration therapy — This group will receive a combined program of conventional physical therapy (30 minutes) and sensory integration therapy (40 minutes) twice weekly for eight weeks (16 sessions, 70 minutes each). Sessions include a warm-up, active phase, and cool-down. Sensory integration therapy targets proprioceptive, visual, and vestibular inputs through progressively challenging balance and gait exercises under varied sensory conditions (eyes open/closed, firm or compliant surfaces), incorporating external and internal perturbations and barefoot gait training, with difficulty individualized and rest provided to prevent fatigue.
  Arms: Conventional physical therapy program + Sensory integration therapy

SUMMARY:
This study aims to evaluate the impact of sensory integration therapy on individuals with multiple sclerosis (MS) by examining its effects on gait variability and overall quality of life.

DETAILED DESCRIPTION:
Rehabilitation interventions within the neurorehabilitation domain (e.g. physiotherapy) have been shown to be beneficial in improving gait disorders in MS, functioning and QoL despite progression of MS. Several systematic reviews report on evidence of rehabilitation in general as well as on specific modalities, e.g. exercise. Therefore, development of affordable and convenient rehabilitation strategies must be emphasized.

Studies report that sensory dysfunctions in patients with multiple sclerosis primarily play a key role in disrupting motor control and mobility including gait abnormalities, reduced balance, altered alignment, range of motion, and coordination. Only a handful of studies have analyzed the effects of external sensory stimulations (auditory, visual) on motor performance in patients with multiple sclerosis. Sensory inputs are a necessary component for motor control and movement performance. Interaction among somatosensory, visual, and vestibular systems is essential for normal motor responses, balance control and mobility. Up to knowledge, there are lack of studies that investigate the effect of sensory integration therapy program on gait variability and quality of life in patients with Multiple Sclerosis. A study states that sensory integration therapy improves a children's capacity to analyze and integrate sensory data by incorporating various visual processing, kinesthetic awareness, tactile awareness, visuomotor coordination development, vestibular and proprioceptive activities. The goal of sensory integration therapy (SIT) is to improve the individual ability to integrate sensory information by strengthening each of the sensory systems (vestibular, proprioception and visual systems).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients diagnosed with MS of relapsing-remitting at least 1 year before this study.
* The Patient's age will range from 18-45.
* A stable MS disease without any episodes of relapse within three months before the study.
* The Expanded Disability Status Scale (EDSS) scale from medical documentation (2-4.5) involve that patients have (visual, cerebellum, pyramidal brainstem and sensory) problems.
* Ability to walk six minutes' walk test (6 min walk test)

Exclusion Criteria:

* Orthopedic disorders such as contracture deformities that could negatively affect gait.
* Other disorders affect gait and quality of life as (diabetes mellitus).
* Other diseases that affect Visual and vestibular problems system (such as vestibular neuritis).
* Marked spasticity grade (2,3,4) for bilateral lower extremities according to modified ashworth scale.
* Pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-07-05 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Step Length Variability | 20 weeks
  Step length variability will be assessed using the Biodex Gait Trainer 2 TM system. Participants will walk on the treadmill at a self-selected comfortable pace for three minutes after a familiarization period of 3-5 minutes. Three successive trials will be conducted with 2-3 minutes rest between trials, and the average will be calculated. Lower coefficient of variance (CV) values indicate less gait variability and better gait stability.
Step cycle Variability | 20 weeks
  Step cycle variability will be measured during continuous walking on the Biodex Gait Trainer 2 TM system. Following familiarization, participants will walk at a comfortable self-selected speed for three minutes. Three trials will be-performed with rest periods in between, and the average CV will be recorded. This measure reflects temporal gait consistency.
Walking Speed Variability | 20 weeks
  Walking speed variability will be evaluated using the Biodex Gait Trainer 2 TM system. After familiarization, participants will walk continuously for three minutes at their comfortable self-selected pace. Three successive trials will be conducted with rest intervals between trials, and the average CV will be recorded to assess speed consistency during walking.
Single Support Time Variability (Time on Each Foot) | 20 weeks
  Single support time (time spent on each foot during walking) variability will be assessed using the Biodex Gait Trainer 2 TM system. Following familiarization with the treadmill, participants will walk at comfortable speed for three minutes. Three trials will be performed with rest periods between trials, and the average CV will be calculated to evaluate single limb stance stability during gait.
Step Length Variability (Smartphone-Based Assessment) | 20 weeks
  Step length will be assessed using a validated smartphone application with the device secured to the participant's third lumbar vertebra (L3-L5 level) using a waist band. Participants will walk along a 7-meter walkway. The smartphone's built-in sensors (accelerometer and gyroscope) will automatically record and calculate step length based on movement patterns.
Gait Velocity Variability (Smartphone-Based Assessment) | 20 weeks
  Walking speed will be measured using a smartphone application validated for gait analysis. The smartphone will be positioned at the lumbar spine (L3-L5) using a secure waist band. Participants will complete walking trials over a 7 meter walkway (two trials). The application will automatically calculate walking speed from sensor data collected during each trial.
Step Time Variability (Smartphone-Based Assessment) | 20 weeks
  Step time will be assessed using a smartphone-based gait analysis application with the device fixed to the participant's lower lumbar region (L3-L5 vertebral level) via waist band. Following the researcher's "start" command, participants will walk along a 7-meter pathway (two trials). The smartphone's sensors will automatically detect and measure the time taken to complete each stride cycle. asked to answer items referring to the activities past 4 weeks. Items within subscales will be totaled to provide a summed score for each subscale or dimension. The responses will be scored in standardized fashion and will be scaled from 0 to 100, where (0= represent the poorest health and 100= represent the best health) in each category. Each subscale can be used independently.
Timed 25 foot walk test | 20 weeks
  The Timed 25-Foot Walk (T25FW) test will be used to assess lower-limb function by measuring the time required to walk 25 feet (7.5 m) as quickly and safely as possible. Patients will perform two trials, and the mean time will be recorded using a stopwatch. Walking speed will be calculated by dividing the distance by the average time, following standardized administration and safety procedures.

SECONDARY OUTCOMES:
Short-form 36 quality of life's (SF-36) | 20 weeks
  The patients will sit in a comfortable relaxed position. The patients will be asked to answer items referring to the activities past 4 weeks. Items within subscales will be totaled to provide a summed score for each subscale or dimension. The responses will be scored in standardized fashion and will be scaled from 0 to 100, where (0= represent the poorest health and 100= represent the best health) in each category. Each subscale can be used independently.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Abo Bakr Elwishy, PhD, Study Chair — Professor, Cairo University; Hossam Mohammed AlSaid, PhD, Study Director — Lecturer, Cairo University
Locations (1):
- Kasr Al Ainy Multiple Sclerosis Clinic, Giza, Egypt